CLINICAL TRIAL: NCT04717414
Title: A Phase 3, Double-blind, Randomized Study to Compare the Efficacy and Safety of Luspatercept (ACE-536) Versus Placebo in Subjects With Myeloproliferative Neoplasm-Associated Myelofibrosis on Concomitant JAK Inhibitor Therapy and Who Require Red Blood Cell Transfusions
Brief Title: An Efficacy and Safety Study of Luspatercept (ACE-536) Versus Placebo in Subjects With Myeloproliferative Neoplasm-Associated Myelofibrosis on Concomitant JAK2 Inhibitor Therapy and Who Require Red Blood Cell Transfusions
Acronym: INDEPENDENCE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACE-536-MF-002; 2020-000607-36 (EudraCT Number); U1111-1260-9595 (Registry Identifier: WHO)
Record Dates: First submitted 2020-12-29; First posted 2021-01-22 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Myeloproliferative Disorders; Myelofibrosis; Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Anemia
Keywords: Luspatercept; ACE-536; Myeloproliferative Neoplasm; Myelofibrosis; JAK2; Red blood cell transfusion; Post-ET MF; Post-PV MF; Reblozyl; Anemia
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Anemia | interventions — luspatercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: Luspatercept (ACE-536) (Experimental): Luspatercept will be given to participants via subcutaneous injection (administered on Day 1 of each 21-day treatment cycle)
  Interventions: Drug: ACE-536
- Control Arm: Placebo (Placebo Comparator): Placebo starting dose with volume equivalent to experimental arm subcutaneous injection every 3 weeks (administered on Day 1 of each 21-day treatment cycle)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ACE-536 — Subcutaneous Injection
  Other Names: Luspatercept; BMS-986346
  Arms: Experimental Arm: Luspatercept (ACE-536)
Other: Placebo — Subcutaneous Injection
  Arms: Control Arm: Placebo

SUMMARY:
The purpose of this Phase 3 study is to evaluate the efficacy and safety of Luspatercept compared with placebo in subjects with myeloproliferative neoplasm (MPN)-associated Myelofibrosis (MF) and anemia on concomitant Janus kinase 2 (JAK2) inhibitor therapy and who require red blood cell count (RBC) transfusions.

The study is divided into Screening Period, a Treatment Phase (consisting of a Blinded Core Treatment Period, a Day 169 Response Assessment, a Blinded Extension Treatment Period, and an Open-label Extension Treatment Period), and a Posttreatment Follow-up Period.

Following the Day 169 Response Assessment, subjects who did not show clinical benefit will have the option to unblind. Subjects who were on placebo during the Blinded Core Treatment Period will have the opportunity to crossover into the Open-Label Extension Treatment Period and receive Luspatercept.

DETAILED DESCRIPTION:
Permitted Concomitant Medications and Procedures

* Subjects are receiving a JAK2 inhibitor for the treatment of MPN-associated MF that is approved in the country where the study is being conducted. JAK2 inhibitors are to be used according to their respective label and as prescribed as part of the subject's standard-of-care therapy as prescribed by their physician prior to study entry.
* Best supportive care (BSC) includes, but is not limited to, treatment with transfusions (eg, RBC, platelet, whole blood), ICTs, antibiotic, antiviral and/or antifungal therapy, and nutritional support as needed.
* Granulocyte colony-stimulating factors (ie, G-CSF, granulocyte macrophage colony-stimulating factor [GM-CSF]) are allowed only in cases of neutropenic fever or as clinically indicated per product label.
* Prophylactic antithrombotic therapy is permitted.
* Thrombopoietin and platelet transfusions are permitted.
* Treatment with systemic corticosteroids is permitted for nonhematological conditions providing the subject is receiving a constant dose equivalent to ≤ 10 mg prednisone during the study.
* Administration of attenuated vaccines (eg, influenza vaccine) is allowed if clinically indicated per Investigator discretion.
* Iron chelation therapy (ICT) is to be used according to the product label. If the label permits, the ICT dose should be stable during at least the first 24 weeks of IP. Initiation of ICT while within the first 24 weeks of IP should be clinically indicated to treat an AE.

Prohibited Concomitant Medications

The following concomitant medications are specifically excluded during the course of study treatment:

* Cytotoxic, chemotherapeutic, targeted, or investigational agents/therapies (excluding JAK2 inhibitor therapy)
* Azacitidine, decitabine, or other hypomethylating agents
* Lenalidomide, thalidomide, and pomalidomide
* Erythropoietin stimulating agents (ESAs) and other RBC hematopoietic growth factors (eg, IL-3)
* Hydroxyurea or other alkylating agents
* Androgens (unless given to treat hypogonadism)
* Oral retinoids (topical retinoids are permitted)
* Arsenic trioxide
* Interferon
* Anagrelide
* Systemic corticosteroids at a dose equivalent to > 10 mg prednisone
* Investigational products for the treatment of MPN-associated MF

ELIGIBILITY:
Subjects must satisfy the following criteria to be randomized in the study:

Inclusion Criteria

- Subject is ≥18 years of age at the time of signing the ICF.

* Subject has a diagnosis of PMF according to the 2016 World Health Organization (WHO) criteria or diagnosis of post-ET or post-PV MF according to the IWG-MRT 2007 criteria, confirmed by the most recent local pathology report.
* Subject is requiring RBC transfusions as defined as:.

  i) Average RBC-transfusion frequency: 4 to 12 RBC units/12 weeks immediately up to randomization. There must be no interval > 6 weeks (42 days) without ≥ 1 RBC transfusion.

ii) RBC transfusions are scored in determining eligibility when given for treatment of:.

A. Symptomatic (ie, fatigue or shortness of breath) anemia with a pretransfusion Hgb ≤ 9.5 g/dL or.

B. Asymptomatic anemia with a pretransfusion Hgb ≤ 7 g/dL.

iii) RBC transfusions given for worsening of anemia due to bleeding or infections are not scored in determining eligibility.

- Subjects on continuous (eg, absent of dose interruptions lasting ≥ 2 consecutive weeks) JAK2 inhibitor therapy as approved in the country of the study site for the treatment for MPN-associated MF as part of their standard-of-care therapy for at least 32 weeks, on stable daily dose for at least 16 weeks immediately up to the date of randomization and anticipated to be on a stable daily dose of that JAK2 inhibitor for at least 24 weeks after randomization.

* Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2.
* A female of childbearing potential (FCBP) for this study is defined as a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (eg, has had menses at any time in the preceding 24 consecutive months). Females of childbearing potential (FCBP)participating in the study must:.

  i) Have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the study, and after end of IP. This applies even if the subject practices true abstinence* from heterosexual contact.

ii) Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, effective contraception** without interruption, 28 days prior to starting IP, during the study therapy (including dose interruptions), and for 12 weeks (approximately 5 times the mean terminal half-life of IP based on multiple-dose PK data) after discontinuation of study therapy.

- Male subjects must: Practice true abstinence* (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential** while participating in the study, during dose interruptions and for at least 12 weeks (approximately 5 times the mean terminal half-life of IP based on multiple-dose PK data) following IP discontinuation, even if he has undergone a successful vasectomy.

i) True abstinence is acceptable when it is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.].

ii) Agreement to use highly effective methods of contraception that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly throughout the course of the study. Such methods include: Combined (estrogen and progestogen containing) hormonal contraception: Oral, Intravaginal, Transdermal; Progestogen-only hormonal contraception associated with inhibition of ovulation: Oral, Injectable hormonal contraception, Implantable hormonal contraception; Placement of an intrauterine device (IUD); Placement of an intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomized partner; Sexual Abstinence.

* Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
* Subject is willing and able to adhere to the study visit schedule and other protocol requirements including the use of the electronic patient reported outcomes device.

Exclusion Criteria

* The presence of any of the following will exclude a subject from randomization:.
* Subject with anemia from cause other than MPN-associated MForJAK2 inhibitor therapy (eg, iron deficiency, vitamin B12 and/or folate deficiencies, autoimmune or hemolytic anemia, infection, or any type of known clinically significant bleeding or sequestration).
* Subject use of hydroxyurea, immunomodulatory compounds such as pomalidomide, thalidomide, ESAs, androgenic steroids or other drugs with potential effects on hematopoiesis ≤ 8 weeks immediately up to the date of randomization.

  i) Systemic corticosteroids are permitted for nonhematological conditions providing the subject is receiving a constant dose equivalent to ≤ 10 mg prednisone for the 4 weeks immediately up to randomization.

ii) Iron chelation therapy (ICT) is permitted providing the subject is receiving a stable dose for the 8 weeks immediately up to randomization.

- Subject with any of the following laboratory abnormalities at screening:.

i) Neutrophils: < 1 x 10^9/L.

ii) White blood count (WBC): > 100 x 10^9/L.

iii) Platelets: the lowest allowable level as approved for the concomitant JAK2 inhibitor but not < 25 x 10^9/L or > 1000 x 10^9/L.

iv) Peripheral blood myeloblasts:> 5%.

v) Estimated glomerular filtration rate:< 30 mL/min/1.73 m2 (via the 4-variable modification of diet in renal disease [MDRD] formula) or nephrotic subjects (eg, urine albumin-to-creatinine ratio > 3500 mg/g).

vi) Aspartate aminotransferase (AST) or alanine aminotransferase (ALT):> 3.0 x upper limit of normal (ULN).

vii) Direct bilirubin: ≥ 2 x ULN.

A. Higher levels are acceptable if these can be attributed to active red blood cell precursor destruction within the bone marrow (eg, ineffective erythropoiesis).

* Subject with uncontrolled hypertension, defined as repeated elevations of systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, that is not resolved at the time of randomization.
* Subject with prior history of malignancies, other than disease under study, unless the subject has been free of the disease for ≥ 3 years. However, subject with the following history/concurrent conditions is allowed:.

  i) Basal or squamous cell carcinoma of the skin.

ii) Carcinoma in situ of the cervix.

iii) Carcinoma in situ of the breast.

iv) Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system).

* Subject with prior hematopoietic cell transplant or subject anticipated to receive a hematopoietic cell transplant during the 24 weeks from the date of randomization. 7. Subject with stroke, myocardial infarction, deep venous thrombosis, pulmonary or arterial embolism within 6 months immediately up to the date of randomization.
* Subject with major surgery within 2 months up to the date of randomization. Subject must have completely recovered from any previous surgery immediately up to the date of randomization.
* Subject with a major bleeding event (defined as symptomatic bleeding in a critical area or organ and/or bleeding causing a decrease in Hgb of ≥ 2 g/dL or leading to transfusion of ≥ 2 units of packed red cells) in the last 6 months prior to the date of randomization.
* Subject with inadequately controlled heart disease and/or have a known left ventricular ejection fraction < 35%.
* Subject with uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
* Subject with known human immunodeficiency virus (HIV), evidence of active Hepatitis B (HepB) as demonstrated by the presence of Hepatitis B surface antigen (HBsAg) and/or positive for Hepatitis B virus DNA (HBVDNA-positive), and/or evidence of active Hepatitis C (HepC) as demonstrated by a positive Hepatitis C virus RNA (HCV-RNA) test of sufficient sensitivity.
* Subject with prior therapy of luspatercept or sotatercept.
* Subject with history of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational product.
* Pregnant or breastfeeding females.
* Subject participation in any other clinical protocol or investigational trial that involves use of experimental therapy (including investigational agents) and/or therapeutic devices within 30 days or for investigational agents within five half-lives, whichever comes later, immediately up to the date of randomization.
* Subject with any significant medical condition, laboratory abnormality, psychiatric illness, or is considered vulnerable by local regulations (eg, imprisoned or institutionalized) that would prevent the subject from participating in the study or places the subject at unacceptable risk if he/she were to participate in the study. 18.Subject with any condition or concomitant medication that confounds the ability to interpret data from the study.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2032-08-18 (Estimated)

PRIMARY OUTCOMES:
Red blood cell-transfusion independence (RBC-TI) ≥ 12 weeks (RBC-TI 12) | Up to 24 weeks
  Proportion of subjects who become RBC-transfusion free over any consecutive 12-week period starting within the first 24 weeks.

SECONDARY OUTCOMES:
Red blood cell-transfusion independence ≥ 16 weeks (RBC-TI 16) | Up to 24 weeks
  Proportion of subjects who become RBC-transfusion free over any consecutive 16-week period
Duration of Red blood cell-transfusion independence (RBC-TI 12) | Up to end of treatment, approximately 3 years
  Maximum duration of RBC-TI response
Reduction of transfusion burden by ≥ 50% and by ≥ 4 units/12 weeks from baseline over any consecutive 12-week period | Up to 24 weeks
  Proportion of subjects who reduce their transfusion burden by ≥ 50% and by ≥ 4 units/12 weeks from baseline over any consecutive 12-week period
Duration of reduction in transfusion burden | Up to end of treatment, approximately 3 years
  Maximum duration of when RBC-transfusion dependent subjects who reduce their transfusion burden by ≥ 50% and by ≥ 4 units/12 weeks from baseline over any consecutive 12 week period
Red blood cell-transfusion independence ≥ 12 weeks in the treatment period (RBC-TI 12/TP) | Up to end of treatment, approximately 3 years
  Proportion of subjects who become RBC-transfusion free over any consecutive 12-week period
Red blood cell-transfusion independence ≥ 16 weeks in the treatment period (RBC-TI 16/TP) | Up to end of treatment, approximately 3 years
  Proportion of subjects who become RBC-transfusion free over any consecutive 16-week period
Change in RBC transfusion burden | Up to 24 weeks
  Mean change in transfusion burden (RBC units) from baseline
Cumulative duration of RBC-transfusion independence | Up to end of treatment, approximately 3 years
  Cumulative response duration for subjects achieving multiple episodes of RBC-TI 12
Mean Hgb increase ≥ 1 g/dL from baseline over any consecutive 12-week period in absence of RBC transfusions | Up to end of treatment, approximately 3 years
  Proportion of subjects achieving a mean Hgb increase ≥ 1 g/dL from baseline over any consecutive 12-week period in absence of RBC transfusions
Change in serum ferritin from baseline | Up to end of treatment, approximately 3 years
  Change in serum ferritin
Incidence of Adverse Events (AEs) | From screening up to 42 days post last dose
  Number of participants with adverse events
Transformation to blast phase: Number of subjects who transform into AML | Up to approximately 5 years
  AML = acute myeloid leukemia
Frequency of Antidrug antibodies (ADA) | From randomization and up to including 48 weeks post first dose
  Will be collected for assessment of anti-drug antibodies (ADA) against Luspatercept in serum in all subjects
Pharmacokinetics - Area Under the Concentration-Time Curve (AUC) | From randomization and up to including 48 weeks post first dose
  Measures of luspatercept exposure area under the curve
Pharmacokinetics - Maximum plasma concentration of drug (Cmax) | From randomization and up to including 48 weeks post first dose
  Maximum plasma concentration of drug

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (185):
- United States (14):
  - Local Institution - 110, Los Angeles, California
  - Local Institution - 135, Orlando, Florida
  - Local Institution - 133, Plantation, Florida
  - Local Institution - 112, Chicago, Illinois
  - Local Institution - 124, Lexington, Kentucky
  - Local Institution - 114, Ann Arbor, Michigan
  - Local Institution - 108, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Local Institution - 130, Knoxville, Tennessee
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Local Institution - 119, Salt Lake City, Utah
- Argentina (3):
  - Local Institution - 172, Ciudad Autónoma de BuenosAires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
- Australia (5):
  - Monash Medical Centre, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Gosford Hospital, Gosford
  - Royal Hobart Hospital, Hobart
- Austria (4):
  - Local Institution - 272, Graz
  - Krankenhaus der Elisabethinen Linz, I Interne Abteilung, Linz
  - Local Institution - 271, Vienna
  - Local Institution - 274, Vienna
- Belgium (8):
  - Local Institution - 318, Bruges
  - Local Institution - 312, Brussels
  - Local Institution - 313, Hasselt
  - Uz Leuven, Leuven
  - Local Institution - 319, Liège
  - Local Institution - 316, Roeselare
  - Local Institution - 315, Verviers
  - Cliniques Universitaires UCL de Mont-Godine, Yvoir
- Canada (8):
  - Local Institution - 181, Calgary, Alberta
  - Local Institution - 179, Edmonton, Alberta
  - Local Institution - 183, Vancouver, British Columbia
  - University Hospital - London Health Sciences Centre, London, Ontario
  - Local Institution - 180, Toronto, Ontario
  - Local Institution - 177, Montreal, Quebec
  - Sir Mortimer B. Davis - Jewish Genl, Montreal, Quebec
  - Local Institution - 176, Sherbrooke, Quebec
- Chile (3):
  - IC La Serena Research, La Serena, Coquimbo Region
  - Local Institution - 192, Las Condes, Metropolitana de Santiago
  - Local Institution - 193, Santiago
- China (20):
  - Nanfang Hospital of Southern Medical University, Guangzhou, GD
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - Local Institution - 804, Nanjing, Jiangsu
  - Local Institution - 818, Nantong, Jiangsu
  - Local Institution - 820, Nanchang, Jiangxi
  - Nanchang University - The Second Affiliated Hospital, Nanchang, Jiangxi
  - Local Institution - 821, Qingdao, Shandong
  - Local Institution - 816, Taiyuan, Shanxi
  - The Second Affiliated Hospital Of Kunming Medical University, Kunming, Yunnan
  - Beijing Peking Union Medical College Hospital, Beijing
  - Local Institution - 802, Changchun
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital Of Harbin Medical University, Harbin
  - Local Institution - 809, Shanghai
  - Local Institution - 801, Shanghai
  - Local Institution - 811, Suzhou
  - Local Institution - 800, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Local Institution - 810, Zhengzhou
- Colombia (3):
  - Local Institution - 161, Medellín, Antioquia
  - Local Institution - 163, Bogotá, Distrito Capital de Bogotai
  - Local Institution - 162, Floridablanca, Soto
- Local Institution - 341, Prague, Czechia
- France (13):
  - Local Institution - 331, Angers
  - Local Institution - 333, Clermont-Ferrand
  - Local Institution - 324, Créteil
  - Chu De Grenoble, Grenoble
  - Local Institution - 327, Lille
  - Local Institution - 332, Lyon
  - CHU de Nice Archet I, Nice
  - Centre Hospitalier Universitaire de Nimes (CHU) - Hopital Universitaire Caremeau, Nîmes
  - Hopital Saint Louis, Paris
  - Groupe Hospitalier Sud Hopital Haut Leveque USN, Pessac
  - CHU La Miletrie, Poitiers
  - ICANS Institut de cancerologie Strasbourg Europe, Strasbourg
  - Local Institution - 330, Toulouse
- Germany (9):
  - Unviversitatsklinikum Aachen, Aachen
  - Stauferklinikum Schwab. Gmund, Baden-Warttemberg
  - Local Institution - 299, Düsseldorf
  - Universitatsklinikum Halle Saale, Halle
  - Local Institution - 300, Hamburg
  - Universitaetsklinikum Jena, Jena
  - Local Institution - 297, Leipzig
  - Local Institution - 301, Mannheim
  - Johannes Wiesling Klinikum Minden, Minden
- Greece (7):
  - Local Institution - 387, Pátrai, Achaia
  - Local Institution - 383, Alexandroupoli
  - Evangelismos General Hospital of Athens, Athens
  - Local Institution - 386, Athens
  - Attikon University General Hospital, Athens
  - University General Hospital of Patras, Rio Patras
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Hong Kong (2):
  - Local Institution - 661, Hong Kong
  - Prince of Wales Hospital the Chinese University of Hong Kong, Shatin
- Hungary (2):
  - Local Institution - 462, Budapest
  - Local Institution - 463, Győr
- Ireland (3):
  - Cork University Hospital, Cork
  - Mater Misercordiae Hospital, Dublin
  - St James Hospital, Dublin
- Israel (5):
  - Tel-Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv
  - Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Shamir Medical Center - Assaf Harofeh, Ẕerifin
- Italy (19):
  - IRCCS - Istituto Romagnolo per lo Studio Dei Tumori "Dino Amadori" (IRST), Meldola (fc), Fc
  - Local Institution - 250, Ancona
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Asst Spedali Civili Di Brescia, Brescia
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele - Ospedale Gaspare Rodolico, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Local Institution - 246, Napoli Campania
  - A.O.U. Maggiore della Carit, Novara
  - Azienda Ospedaliera Di Padova, Padua
  - Local Institution - 248, Pisa
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria
  - Azienda Policlinico Universitario Umberto I, Roma
  - Local Institution - 251, Roma
  - Local Institution - 249, Roma
  - Local Institution - 245, Terni
  - Local Institution - 259, Torino
  - Universita degli Studi dell'Insubria - Ospedale di Circolo e Fondazione Macchi - Varese, Varese
  - Centro Ricerche Cliniche di Verona S.r.l., Verona
- Japan (18):
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki, Nagasaki
  - Kindai University Hospital- Osakasayama Campus, Sayama, Osaka
  - Local Institution - 701, Bunkyo-ku, Tokyo
  - Local Institution - 709, Chūō, Yamanashi
  - Aomori Prefectural Central Hospital, Aomori
  - Local Institution - 713, Bunkyō City
  - Tokai University Hospital, Isehara City, Kanagawa
  - Local Institution - 717, Kamakura
  - Kameda General Hospital, Kamogawa
  - Local Institution - 706, Maebashi
  - University of Miyazaki Hospital, Miyazaki
  - Osaka Metropolitan university Hospital, Osaka
  - Ogaki Municipal Hospital, Ōgaki
  - Local Institution - 708, Sapporo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku
  - Local Institution - 710, Shinjyuku-ku
  - Toyohashi Municipal Hospital, Toyohashi
- Lebanon (3):
  - Local Institution - 551, Saida, South
  - Local Institution - 550, Badaro Beirut
  - Local Institution - 552, Beirut
- Poland (6):
  - Local Institution - 436, Gdansk
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewódzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Local Institution - 433, Poznan
  - Specjalistyczny Szpital im. dra Alfreda Sokolowskiego, Wałbrzych
  - Local Institution - 435, Wroclaw
- Romania (4):
  - Local Institution - 395, Craiova, Dolj
  - Onco Card SRL, Brasov
  - Local Institution - 391, Bucharest
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
- Russia (3):
  - Local Institution - 500, Moscow
  - Local Institution - 503, Saint Petersburg
  - Local Institution - 502, Saint Petersburg
- South Korea (7):
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun-Gun
  - Local Institution - 643, Seongnam-si
  - Local Institution - 647, Seoul
  - The Catholic University of Korea Seoul - Saint Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (11):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol ICO Badalona, Barcelona
  - Local Institution - 208, Granada
  - Hospital Universitario De Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Local Institution - 202, Palma de Mallorca
  - Universitario de Salamanca - Hospital Clinico, Salamanca
  - Complejo Hospitalario Universitario De Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario De Valencia, Valencia
- United Kingdom (4):
  - Nottingham City Hospital, Nottingham, Nottinghamshire
  - Heart of England NHS Foundation Trust, Birmingham
  - United Lincolnshire Hospitals NHS Trust, Boston
  - Churchhill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04717414.html